CLINICAL TRIAL: NCT04357808
Title: Randomized Open Pilot Study to Evaluate the Efficacy of Subcutaneous Sarilumab in Patients With Moderate-severe COVID-19 Infection
Brief Title: Efficacy of Subcutaneous Sarilumab in Hospitalised Patients With Moderate-severe COVID-19 Infection (SARCOVID)
Acronym: SARCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maria del Rosario Garcia de Vicuña Pinedo (Other)
Collaborators: Instituto de Investigación Sanitaria Hospital Universitario de la Princesa (Other)
Responsible Party: Sponsor-Investigator, Maria del Rosario Garcia de Vicuña Pinedo, MD, PhD, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARCOVID; 2020-001634-36 (EudraCT Number)
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Covid-19
Keywords: COVID; SARS-CoV-2; coronavirus infections; sarilumab; IL-6 receptor inhibitors
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sarilumab

STUDY DESIGN:
Intervention Model Description: Randomised, open-label, single-center, comparative trial of sarilumab plus standard of care vs. standard of care in a 2:1 ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sarilumab plus standard of care (Experimental): Sarilumab 200 mg, 2 sc injections in pre-filled syringe or pen, single dose. Treatment with drugs or procedures in routine clinical practice that the clinician responsible for the patient deems necessary is allowed
  Interventions: Drug: Sarilumab
- Standard of care (Active Comparator): Treatment with drugs or procedures in routine clinical practice
  Interventions: Other: Standar of care

INTERVENTIONS:
Drug: Sarilumab — Single dose treatment with sarilumab 2 x 200 mg subcutaneously
  Other Names: Kevzara; SAR153191
  Arms: Sarilumab plus standard of care
Other: Standar of care — Usual clinical care
  Arms: Standard of care

SUMMARY:
The global health emergency created by the rapid spread of the SARS-CoV-2 coronavirus has pushed healthcare services to face unprecedent challenges to properly manage COVID-19 severe and critical manifestations affecting a wide population in a short period of time. Clinicians are committed to do their best with a great uncertainty in this evolving crisis. Off label use of plenty of drugs has arisen the need for clinical trials to demonstrate their true role in the therapy. Based in unpublished experiences in China, Italy and Spain, intravenous IL-6 receptor inhibitors are now being tested in several trials but no data on subcutaneous formulations are available yet. Sarilumab is a human monoclonal antibody that binds membrane-bound and soluble IL-6 receptors to inhibit IL-6 signalling, licensed in a subcutaneous route administration.

DETAILED DESCRIPTION:
SARCOVID is an investigator-initiated monocentric randomised proof of concept study that aims to evaluate the efficacy and safety of a single dose of sarilumab, in subcutaneous administration, in hospitalised patients with moderate to early severe COVID-19 infection, compared to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other validated commercial or public health assay
* Documented interstitial pneumonia requiring admission and at least two of the following:

  1. Fever ≥ 37.8ºC (tympanic)
  2. IL-6 in serum ≥ 25 ng / mL (in the absence of a previous dose of prednisone or equivalent> 1 mg / kg) or PCR> 5mg / dL
  3. Lymphocytes <600 mm3
  4. Ferritin> 300 mcg / L that doubles in 24 hours
  5. Ferritin> 600 mcg / L in the first determination and LDH> 250 U / L
  6. D-dimer (> 1 mg / L)
* Informed verbal or administration consent under urgent conditions, documented in the electronic medical record.

Exclusion Criteria:

* Patients who require mechanical ventilation at the time of inclusion.
* AST / ALT values > 5 folds upper normal limit.
* Neutrophil count below 500 cells / mm3
* Platelet count below 50,000 cells / mm3
* Documented sepsis or high suspicion by pathogens other than COVID-19.
* Presence of comorbidities that according to clinical judgment could lead to an unfavorable result.
* Complicated diverticulitis or intestinal perforation.
* Current skin infection (eg, uncontrolled dermopiodermitis).
* Immunosuppressive anti-rejection therapy.
* Pregnancy or lactation.
* Previous treatment with tocilizumab or sarilumab.
* Patients participating in some other clinical trial for SARS-CoV-2 infection.
* Patients with known hypersensitivity or contraindication to sarilumab or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Mean change in clinical status assessment using the 7-point ordinal scale at day 7 after randomisation | 7 days from enrolment
  Score ranges 1-7
  1. Death;
  2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized
Duration of hospitalisation (days) | 30 days from enrolment
  Days from the date of enrolment to the date of discharge
Death | 30 days from enrolment
  Number of deaths

SECONDARY OUTCOMES:
Time to become afebrile (days) | 30 days from enrolment
  Time to become afebrile for a minimum period of 48 hours, without antipyretics
Time to non-invasive mechanical ventilation (days) | 30 days from enrolment
  Days from enrolment to non-invasive mechanical ventilation
Time to invasive mechanical ventilation (days) | 30 days from enrolment
  Days from enrolment to invasive mechanical ventilation
Time to independence from supplementary oxygen therapy (days) | 30 days from enrolment
  Days from enrolment to supplementary oxygen therapy withdrawal
Mean change in clinical status assessment using the 7-point ordinal scale at day 14 after randomisation | 14 days from enrolment
  Scale ranges 1-7:
  1. Death
  2. Hospitalized, with mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  3. Hospitalized, with non-invasive mechanical ventilation, a mask with a reservoir or oxygen with high flow nasal goggles.
  4. Hospitalized with oxygen supplement
  5. Hospitalized, without oxygen supplement, but in need of continued medical care (related or not with COVID)
  6. Hospitalized, without oxygen supplement and without the need for continued medical care
  7. Not hospitalized

OTHER OUTCOMES:
Incidence of serious and non-serious adverse events. | 30 days after enrolment
  Number of adverse events and number of patients with adverse events
Discontinuation due to adverse reactions | 30 days after enrolment
  Number of adverse reactions that requires discontinuation of any drug in the study

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Garcia de Vicuña, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

REFERENCES:
- [Derived] Garcia-Vicuna R, Rodriguez-Garcia SC, Abad-Santos F, Bautista Hernandez A, Garcia-Fraile L, Barrios Blandino A, Gutierrez Liarte A, Alonso-Perez T, Cardenoso L, Alfranca A, Mejia-Abril G, Sanz Sanz J, Gonzalez-Alvaro I. Subcutaneous IL-6 Inhibitor Sarilumab vs. Standard Care in Hospitalized Patients With Moderate-To-Severe COVID-19: An Open Label Randomized Clinical Trial. Front Med (Lausanne). 2022 Feb 23;9:819621. doi: 10.3389/fmed.2022.819621. eCollection 2022. PMID 35280907
- [Derived] Garcia-Vicuna R, Abad-Santos F, Gonzalez-Alvaro I, Ramos-Lima F, Sanz JS. Subcutaneous Sarilumab in hospitalised patients with moderate-severe COVID-19 infection compared to the standard of care (SARCOVID): a structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Sep 9;21(1):772. doi: 10.1186/s13063-020-04588-5. PMID 32907638